CLINICAL TRIAL: NCT02871037
Title: A Phase 1, 3-part Study Of Pf-05221304 In Healthy Adults: Part 1 - Randomized, Double-blind, Placebo-controlled Assessment Of Safety And Pharmacokinetics Of Single, Escalating, Oral Doses; Part 2 - Randomized, Double-blind, Placebo-controlled Assessment Of Safety And Pharmacokinetics Of Repeated, Escalating, Oral Doses; Conditional Part 3 - Effect Of Food On The Pharmacokinetics Of Pf-05221304
Brief Title: Single Dose, Repeated Dose, and Conditional Food Effect Study of PF-05221304 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Basic Science
Other Study IDs: C1171001
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2018-05-24 (Actual); Status verified 2018-05

CONDITIONS: Normal Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- Part 1_Cohort 1_Active (Experimental): Single, escalating dose of PF-05221304
  Interventions: Drug: PF-05221304
- Part 1_Cohort 1_Placebo (Placebo Comparator): Single dose of Placebo
  Interventions: Other: Placebo
- Part 1_Cohort 2_Active (Experimental): Single, escalating dose of PF-05221304
  Interventions: Drug: PF-05221304
- Part 1_Cohort 2_Placebo (Experimental): Single dose of Placebo
  Interventions: Other: Placebo
- Part 2_Active (Experimental): Repeated, escalating doses of PF-05221304
  Interventions: Drug: PF-05221304
- Part 2_Placebo (Placebo Comparator): Repeated doses of placebo
  Interventions: Other: Placebo
- Part 3 (Experimental): Single dose of PF-05221304 with and without food
  Interventions: Drug: PF-05221304

INTERVENTIONS:
Drug: PF-05221304 — Single or repeated, escalating dose of PF-05221304
  Arms: Part 1_Cohort 1_Active; Part 1_Cohort 2_Active; Part 2_Active; Part 3
Other: Placebo — single or repeated dose of placebo
  Arms: Part 1_Cohort 1_Placebo; Part 1_Cohort 2_Placebo; Part 2_Placebo

SUMMARY:
The current study is the first clinical trial proposed with PF-05221304. It is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) following administration of single and repeated doses of PF-05221304 to healthy adult subjects. The study may also evaluate effect of food on PK of PF-05221304.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and female of non-childbearing potential;
* Body Mass Index 17.5-30.5 kg/m2;
* Body weight >50 kg;

Exclusion Criteria:

* Evidence of history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergises, but excluding untreated, asymptomatic, seasonal allergies at time of dosing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of Subjects experiencing an Adverse Event | Screening up to 28 days after last dose of study medication
  Assessment by adverse event monitoring, 12 lead ECGs, telemetry, vital signs and clinical safety laboratory measurements.
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.
Part 2: Number of Subjects experiencing an Adverse Event | Screening up to 28 days after last dose of study medication
  Assessment by adverse event monitoring, 12 lead ECGs, telemetry, vital signs and clinical safety laboratory measurements.
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.
Part 3: Maximum Observed Plasma Concentration (Cmax) for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Part 3: Time to Reach Maximum Observed Concentration for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Part 3: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Part 3: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  AUC (0-infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Part 3: Plasma Decay Half-Life (t1/2) for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Part 3: Apparent Total Body Clearance (CL/F) for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after apparent total body clearance is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Part 3: Apparent Volume of Distribution (Vz/F) for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

SECONDARY OUTCOMES:
Part 1:Maximum Observed Plasma Concentration (Cmax) for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Maximum Observed Plasma Concentration (Cmax)
Part 1: Time to Reach Maximum Observed Concentration for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Part 1: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast)
Part 1: dose-normalized Cmax and AUClast for PF05221304 | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
Part 1: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0- infinity)] for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  AUC (0-infinity)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Part 1: Plasma Decay Half-Life (t1/2) for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Plasma Decay Half-Life (t1/2)
Part 1: Apparent Total Body Clearance (CL/F) for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after apparent total body clearance is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Part 1: Apparent Volume of Distribution (Vz/F) for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 5, 8, 12, 16, 24, 36, and 48 hours post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Part 2: Single dose plasma parameters of Cmax for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose on Day 1
  Maximum Observed Plasma Concentration (Cmax)
Part 2: Single-dose plasma parameters of Tmax for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose on Day 1
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Part 2: Single-dose plasma parameters of Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau) for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose on Day 1
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau)
Part 2: Multiple-dose plasma parameters of Cmax for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose for Day 7; (and Day 14, as permitted)
  Maximum Observed Plasma Concentration (Cmax)
Part 2: Multiple-dose plasma parameters of Tmax for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose for Day 7; (and Day 14, as permitted)
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Part 2: Multiple-dose plasma parameters of AUCtau for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose for Day 7; (and Day 14, as permitted)
  Area under the concentration curve from time 0 to end of dosing interval (AUCtau)
Part 2: Multiple-dose plasma parameters of Minimum Observed Plasma Trough Concentration (Cmin) for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose for Day 7; (and Day 14, as permitted)
Part 2: Multiple-dose plasma parameters of CL/F for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose for Day 7; (and Day 14, as permitted)
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after apparent total body clearance is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Part 2: Multiple-dose plasma parameters of Vz/F for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours on Day 1 and 7, and 0 hr on Day 2, Day 4, Day 8, Day 10, Day 13, Day 15, and Day 16 post dose
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.
Part 2: Multiple-dose plasma parameters of Peak-trough ratio (PTR) for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose for Day 7; (and Day 14, as permitted)
Part 2: Multiple-dose plasma parameters of Observed accumulation ratio for Cmax (Rac(Cmax)) for PF-05221304 | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose for Day 7; (and Day 14, as permitted)
Part 2: Multiple-dose plasma parameters of Observed accumulation ratio (Rac(AUCtau)) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, and 24 hours post dose for Day 7; (and Day 14, as permitted)
Part 2: Multiple-dose plasma parameters of Plasma Decay Half-Life (t1/2) for PF-05221304 (as permitted) | 0, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, and 16 hours on Day 1 and 7, and 0 hr on Day 2, Day 4, Day 8, Day 10, Day 13, Day 15, and Day 16 post dose
  Plasma Decay Half-Life (t1/2)
Part 3: Number of Subjects experiencing an Adverse Event | Screening up to 28 days after last dose of study medication
  Assessment by adverse event monitoring, 12 lead ECGs, telemetry, vital signs and clinical safety laboratory measurements.
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a subject who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug was assessed by the investigator (Yes/No). Subjects with multiple occurrences of an AE within a category were counted once within the category.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1171001&StudyName=A+Phase+1%2C+3-part+Study+In+Healthy+Adults+%3A+Part+1+%E2%80%93+Randomized%2C+Double-blind%2C+Placebo+Controlled+Assessment+Of+Safety+And+Pharmacokinetics+Of+Single%2C+Escalating%2C+Oral+Doses+Of+Pf+05221304%3B+Part+2+%E2%80%93+Randomized%2C+Double-blind%2C+Placebo+Controlled+Assessment+Of+Safety%2C+And+Pharmacokinetics+Of+Repeated%2C+Escalating%2C+Oral+Doses+Of+Pf+05221304%3B+Part+3+%E2%80%93+Characterization+Of+The+Effect+Of+Food+On+Pharmacokinetics+Of+Pf+05221304
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=C1171001&StudyName=A+Phase+1%2C+3-part+Study+Of+Pf-05221304+In+Healthy+Adults%3A+Part+1+%E2%80%93+Randomized%2C+Double-blind%2C+Placebo-controlled+Assessment+Of+Safety+And+Pharmacokinetics+Of+Single%2C+Escalating%2C+Oral+Doses%3B+Part+2+%E2%80%93+Randomized%2C+Double-blind%2C+Placebo-controlled+Assessment+Of+Safety+And+Pharmacokinetics+Of+Repeated%2C+Escalating%2C+Oral+Doses%3B+Conditional+Part+3+%E2%80%93+Effect+Of+Food+On+The+Pharmacokinetics+Of+Pf-05221304